CLINICAL TRIAL: NCT01376687
Title: Osteopathic Manipulative Medicine and Kinetics
Status: Completed | Type: Observational
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Tamara Reid Bush, Assistant Professor, Michigan State University
Other Study IDs: OMMGLOVE
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Cervical Spine
Keywords: Osteopathic Medicine; Cervical Spine; Kinetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pain free: No pain in the cervical spine
- Pain: Pain of 3 or greater on a VAS scale for the cervical spine

SUMMARY:
Back pain affects the majority of the population at some time. Currently there are no published and scientifically accepted objective measures to support manual medicine diagnostic and treatment techniques for back pain. The purpose of this project is to collect and evaluate objective (pressure and motion) data from standard clinical diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* HEalthy and no pain in cervical spine
* Pain of 3 or greater in cervical spine

Exclusion Criteria:

* pain of less than 3 in the cervical spine region
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HEalthy and no pain in cervical spine Pain of 3 or greater in cervical spine
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of obtaining force data during clinical assessment | 1 year
  Assessment of force sensing equipment while conducting clinical diagnoses

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States